CLINICAL TRIAL: NCT05764200
Title: Acute Microbial Switch Study
Brief Title: Acute Microbial Switch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL82078.068.22
Record Dates: First submitted 2023-02-17; First posted 2023-03-10 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Insulin Sensitivity; Glucose Metabolism Disorders (Including Diabetes Mellitus); Hyperinsulinism
Keywords: microbiota; insulin sensitivity; fiber
MeSH Terms: conditions — Insulin Resistance; Glucose Metabolism Disorders; Hyperinsulinism

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lean normoglycaemic individuals fiber mixture (Active Comparator): Two day supplementation of 12 g (3 x 4 g) of the dietary fiber inulin in combination with 9.375 g (3 x 3.125 g (80% resistant starch (3 x 2.5 g)) granular potato starch
  Interventions: Dietary Supplement: Two day supplementation of a complex fiber mixture
- lean normoglycaemic placebo (Placebo Comparator): Two day supplementation of 11.43 g (3 x 3.81 g) maltodextrin
  Interventions: Dietary Supplement: Placebo supplementation
- overweight and/or obesity and prediabetes/insulin fiber mixture (Active Comparator): Two day supplementation of 12 g (3 x 4 g) of the dietary fiber inulin in combination with 9.375 g (3 x 3.125 g (80% resistant starch (3 x 2.5 g)) granular potato starch
  Interventions: Dietary Supplement: Two day supplementation of a complex fiber mixture
- overweight and/or obesity and prediabetes/insulin resistance placebo (Placebo Comparator): Two day supplementation of 11.43 g (3 x 3.81 g) maltodextrin
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Two day supplementation of a complex fiber mixture — Participants will undergo a two day supplementation of a complex fiber supplement vs. placebo with a two-week washout period between the two interventions in a randomized order
  Arms: lean normoglycaemic individuals fiber mixture; overweight and/or obesity and prediabetes/insulin fiber mixture
Dietary Supplement: Placebo supplementation — Participants will undergo a two day supplementation of a complex fiber supplement vs. placebo with a two-week washout period between the two interventions in a randomized order
  Arms: lean normoglycaemic placebo; overweight and/or obesity and prediabetes/insulin resistance placebo

SUMMARY:
In this project the investigators will test if it is possible to measure changes in intestinal gas production after supplementation of a complex fiber mixture over a 36 hour period in both lean normoglycemic individuals and individuals with insulin resistance and/or prediabetes with overweight when compared with a placebo

Changes in intestinal gas production will also be related to energy expenditure, substrate metabolism, microbial composition and related metabolites in feces, blood and urine.

DETAILED DESCRIPTION:
In this project the investigators aim to test whether it is possible to precisely measure the changes in fermentation gas patterns after supplementation of a complex fibre mixture over a 36-hour period in both lean normoglycemic and individuals with insulin resistance and/or prediabetes with overweight when compared with a placebo. Additionally, the investigators will investigate whether changes in fermentation patterns will be directly related to changes in carbohydrate and fat oxidation and to microbial composition or related metabolites and hormones in blood, faeces, and urine.

ELIGIBILITY:
Inclusion Criteria:

* Lean normoglycemic individuals:
* Lean (BMI ≥ 18.5 kg/m2 and ≤ 24.9 kg/m2 );
* Normal fasting glucose (plasma glucose < 5.6 mmol/L) and a HOMA-IR< 2.2

Individuals with overweight/obesity and prediabetes/insulin resistance:

* Overweight/obesity (BMI ≥ 28 kg/m2 and ≤ 40 kg/m2 );
* insulin resistance (HOMA-IR>2.2) and/or impaired fasting glucose (IFG: plasma glucose ≥ 5.6 mmol/l)

For both subject groups:

* Aged 30 - 75 years;
* Normal blood pressure (systolic blood pressure 100-150mmHg, diastolic blood pressure 60-100 mmHg);
* Weight stable for at least 3 months (± 2 kg)

Exclusion Criteria:

* T2DM (defined as fasting plasma glucose ≥ 7.0 mmol/L)
* Gastroenterological diseases
* Abdominal surgery affecting the GI tract;
* Cardiovascular diseases, cancer, liver or kidney malfunction, disease with a life expectancy shorter than five years;
* Abuse of products;

  * Alcohol (> 15 standard units per week)
  * Drugs
  * Excessive nicotine use defined as >20 cigarettes per day;
* Plans to lose weight or following of a hypocaloric diet
* Regular supplementation of pre- or probiotic products, use of pre- or probiotics three months prior to the start of the study;
* Intensive exercise training more than three hours a week;
* Use of most medications that influence glucose or fat metabolism, like some lipid lowering-drugs (e.g., PPAR γ or PPARα (fibrates) agonists), glucose-lowering agents (including all sulfonylureas, biguanides, α-glucosidase inhibitors, thiazolidinediones, repaglinide, nateglinide and insulin), inflammation (e.g., anti-inflammatory* or immunosuppressive drugs) and anti-oxidants;
* Regular use of laxatives;
* Use of antibiotics in the last three months (antibiotics use can alter substantially the gut microbiota composition).
* Veganism
* Lactose intolerance
* For women: pregnancy or lactation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
24 hour intestinal gas concentrations | after ingestion of the supplement up until 24 hours after supplementation continuously
  changes in intestinal gas excretion (methane, hydrogen or hydrogen sulphide will be measured using gas sensors in a modified respiration chamber)

SECONDARY OUTCOMES:
24 hour energy expenditure | after ingestion of the supplement up until 24 hours after supplementation continuously
  changes in 24 hour energy expenditure will be measured in a respiration chamber
24 hour substrate metabolism | after ingestion of the supplement up until 24 hours after supplementation continuously
  changes in 24 hour substrate metabolism will be measured in a respiration chamber (fat and carbohydrate oxidation)
fecal microbial metabolite concentrations | after ingestion of the supplement and 24 hours after supplementation
  the concentrations of fecal SCFA and BCFAs will be measured
Fecal microbiota composition | at baseline and 24 hours after supplementation
  Faecal microbiota composition will be assessed via16S rRNA gene sequencing
24 hour glucose monitoring | after ingestion of the supplement up until 24 hours after supplementation
  24 hour glucoses concentrations will be measured using a wearable monitor during each testday
circulating blood markers | after ingestion of the supplement at multiple timepoints up until 24 hours after supplementation
  plasma blood glucose, insulin, GLP-1, glucagon, PYY, triglycerides, FFA, SCFA and BCFA
Urine metabolites | at baseline up until 24 hours after supplementation
  urinary concentrations of phenolic compounds, p-cresol and nitrogen will be measured

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Department of Human Biology, Maastricht University Medical Centre, Maastricht
  - Maastricht University Medical Centre, Maastricht

IPD SHARING:
Plan to Share IPD: Undecided
anonymized data may be shared with other researchers for meta-analyses etc., however personalized data names etc. will not be made available